CLINICAL TRIAL: NCT00770406
Title: Intravesikal Instillation af Botulinum Toxin Type A Til Patienter Med Urge Urininkontinens
Brief Title: Intravesical Instillation of Botulinum Toxin Type A to Patients With Urge Urinary Incontinence
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Soren Brostrom, MD, PhD, Glostrup University Hospital,Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTXA2008
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Urge Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: botulinum toxin type A — 100 or 200 units intravesically

SUMMARY:
A pilot study to examine efficacy and safety of intravesical botulinum toxin type A.

ELIGIBILITY:
Inclusion Criteria:

* refractory urge urinary incontinence

Exclusion Criteria:

* neurological disease
* pregnant or lactating
* bladder neoplasias

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Incontinence episode frequency | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Copenhagen, Denmark